CLINICAL TRIAL: NCT01266746
Title: Clinical Observation of Postoperative Status of Macular Hole in Gas-filled Eyes by Spectral Domain-optical Coherence Tomography
Brief Title: Optical Coherence Tomography in Gas-filled Eyes
Status: Completed | Type: Observational
Sponsor: Kyorin University (Other)
Responsible Party: Principal Investigator, Makoto Inoue, Associate professor, Kyorin University
Other Study IDs: Kyorineye001; KYORIN-H21012 (Other: Kyorin University School of Medicine)
Record Dates: First submitted 2010-12-20; First posted 2010-12-24 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2012-12

CONDITIONS: Macular Hole
Keywords: gas tamponade,; macular hole,; macular hole retinal detachment,; optical coherence tomography
MeSH Terms: conditions — Retinal Perforations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Macular hole: The patients of idiopathic macular hole enrolled in the study
  Interventions: Procedure: Vitreous surgery
- Macular hole retinal detachment: The patients of macular hole retinal detachment enrolled in the study
  Interventions: Procedure: Vitreous surgery
- Myopic traction maculopathy: The patients of macular hole with myopic traction maculopathy enrolled in the study
  Interventions: Procedure: Vitreous surgery

INTERVENTIONS:
Procedure: Vitreous surgery — Vitreous surgery is performed to treat the original disease not for the study.

SUMMARY:
The aim of this study is to determine the condition to detect the status of a macular hole by spectral domain optical coherence tomography (SD-OCT) in gas-filled eyes. The macular area is scanned by SD-OCT (OCT-4000, Carl Zeiss Meditec) in the patients who underwent vitreous surgery for macular hole to detect macular jole closure on postoperative days 1, 3, 7, and 30.

DETAILED DESCRIPTION:
We studied 26 eyes with an idiopathic macular hole (MH), 7 eyes with a MH retinal detachment (MHRD), and 4 eyes with a MH with myopic traction maculopathy. This was a prospective study conducted between April 2009 and August 2009 at the Kyorin Eye Center of the Kyorin University School of Medicine, Tokyo, Japan. The age, gender, laterality of the diseased eye, stage of MH based on the Gass classification, and Snellen best-corrected visual acuity (BCVA) were recorded. The axial length was measured with the OA1000 (TOMEY Corp., Nagoya, Japan) preoperatively in eyes with MH and postoperatively in eyes with MHRD and myopic traction maculopathy to avoid the effect of retinal detachment on the axial length. The presence of a posterior staphyloma within the posterior vascular arcade was determined by ophthalmoscopy and ultrasonography (Ultrascan®, Alcon Laboratories, Fort Worth, TX).

Standard pars plana vitrectomy was performed. The internal limiting membrane (ILM) was removed after making it visible with triamcinolone acetonide (Kenacort-A®, Bristol Pharmaceuticals KK, Tokyo, Japan) or indocyanine green (Santen Pharmacy, Osaka, Japan) in all eyes. Preoperative cataracts were graded as mild (nuclear sclerosis 1+) or moderate to advanced (nuclear sclerosis 2+ or 3+), and phacoemulsification with implantation of an intraocular lens was performed on all cataractous eyes higher than grade 1. Room air, 20% sulfur hexafluoride (SF6), or 14% perfluoropropane (C3F8) was used to tamponade the retina. When the MH was confirmed to be closed in the patients with a idiopathic MH, the face-down position was discontinued although the patients were instructed to avoid an upright position. Patients with MHRD and myopic traction maculopathy were instructed to keep a facedown position for one to two weeks even after a MH closure was detected.

All surgery was performed under retrobulbar anesthesia, and a written informed consent was obtained from all patients after a full explanation of the purpose and possible complications of the treatment. The study protocol was approved by the Institutional Review Committee of the Kyorin University School of Medicine and all of the patients approved the clinical review of their medical records.

The entire macular area was scanned by SD-OCT (OCT4000, Cirrus HD-OCT, Carl Zeiss Medic Inc., Dublin, California, USA) in the sitting position to avoid missing a MH. The 5-line raster mode was used to obtain high quality images on postoperative days 1, 3, 7, and 30. When a macular image could not be obtained, the patients were instructed to look slightly downward or upward until a clearer view of the macular area was obtained in the OCT images. The ability to detect a closed MH or the status of the foveal detachment or schisis by the SD-OCT was evaluated, and the pre- and postoperative factors that affected the OCT images were investigated. The volume of intravitreal gas was estimated by the level of the inferior gas meniscus at the retina with an indirect ophthalmoscope in a sitting position.

ELIGIBILITY:
Inclusion Criteria:

* the patients who had a vitreous surgery for macular hole, macular hole retinal detachment, macular hole with myopic traction maculopathy and examined spectral domain optical coherence tomography preoperatively and postoperatively.

Exclusion Criteria:

* the patients who had vitreous surgery for other disease
* the patients who did not have postoperative examination of spectral domain optical coherence tomography

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients who had a vitreous surgery for macular hole, macular hole retinal detachment, myopic traction maculopathy and examined spectral domain optical coherence tomography preoperatively and postoperatively.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2009-04; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
macular hole closure detected by spectral domain optical coherence tomography | Change from preoperative status up to postoperative day 30.
  The maular hole closure in eyes with intravitreal gas is detected by spectral domain optical coherence tomography

SECONDARY OUTCOMES:
preoperative and postoperative vision | This was a prospective study conducted between April 2009 and August 2009. The vision is measured preoperatively and postoperative day 30.
  The preoperative and postoperarive vision are measured.

CONTACTS AND LOCATIONS:
Overall Officials: Makoto INoue, MD, Principal Investigator — Kyorin Eye Center
Locations (1):
- Kyorin Eye Center, Mitaka, Tokyo, Japan